CLINICAL TRIAL: NCT05810922
Title: Arbutus Berry - Intervention Study to Evaluate the Modulation of Intestinal Microbiota and Metabolic Parameters
Acronym: F4F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Associação Centro de Apoio Tecnológico Agro-Alimentar de Castelo Branco (CATAA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F4F- Forest for Future
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Diet Habit
Keywords: adipokines; arbutus berry; gut microbiota; inflammatory cytokines; short chain fatty acid; strawberry tree
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: one group consuming 50 g of arbutus berry/day one group consuming 200 g of arbutus berry/day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 g arbutus berry (Experimental): consumption of 50 g arbutus berry/day for 14 days
  Interventions: Other: arbutus berry
- 200 g arbutus berry (Experimental): consumption of 200 g arbutus berry/day for 14 days
  Interventions: Other: arbutus berry

INTERVENTIONS:
Other: arbutus berry — consumption of 50 g arbutus berry/day or 200 g arbutus berry/day for 14 days

SUMMARY:
The tree that produces the arbutus berry, the strawberry tree, scientific name Arbutus unedo L., belongs to the family of Ericaceae. It exists in almost all of Southern Europe in arid and siliceous lands, in woods and forests and is very common in Portugal.

Known for its use in the production of liqueurs and brandy, the arbutus berry is a fruit that can be consumed in nature or incorporated in the preparation of other foods. Arbutus berry has been attributed some properties beneficial to health given its low caloric value and its high content of vitamin C and flavonoids, which is why it is considered a good source of antioxidants.

Arbutus has a high carbohydrate content (70-80% dry weight) with a relevant fiber fraction (10-30%), constituting an interesting source of vegetable protein (1-9%) and lipids (2-3%). Given this interesting nutritional composition, the hypothesis is that a daily consumption of this fruit can have an impact in health outcomes such as microbiota modulation and an improvement of metabolic parameters.

DETAILED DESCRIPTION:
The main objective of this clinical trial is to evaluate the effect of including a daily consumption of arbutus berry on the composition and diversity of the intestinal microbiota. It is also intended to evaluate metabolic parameters to determine the impact of this intervention.

Participants will consume 50g or 200g of arbutus berry daily for 4 weeks. This study aims to provide scientific evidence regarding the impact of arbutus berry consumption on intestinal microbiota and general health improvements.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian.
* Age between 18 and 50 years.
* Filling informed consent.
* Body mass index (BMI) between 18,5 kg/m2 and 25 kg/m2.

Exclusion Criteria:

* Arbutus berry sensibility.
* Arbutus berry daily consumption in the month before the study begin.
* Having taken antibiotics within the 6 months prior to beginning the study.
* Use of pro/prebiotics or fiber as a dietary supplement or any food/molecule that modifies intestinal transit time 6 weeks before recruitment.
* Use of laxative 6 weeks before recruitment.
* Specific nutritional therapy (e.g. high protein).
* Excessive alcohol consumption.
* Smoking.
* Diagnosis of gastrointestinal pathology, hormonal or thyroid pathology, autoimmune diseases, chronic use of corticosteroids, psychiatric disease or Diabetes Mellitus.
* Use of proton pump inhibitors, antidiabetic drugs, insulin, or statins.
* Pregnant or breastfeeding.
* Participation in another clinical trial within the last 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota characterization | 14 days
  Difference in gut microbiota taxonomic characterization, from baseline to the end of intervention
Changes in gut microbiota diversity | 14 days
  Difference in gut microbiota Shannon index, from baseline to the end of intervention

SECONDARY OUTCOMES:
Changes in fasting glucose | 14 days
  Changes in fasting glucose, measured in mg/dL, from baseline to end of intervention
Changes in HOMA-IR | 14 days
  Changes in HOMA-IR from baseline to end of intervention
Changes in HDL cholesterol | 14 days
  Changes in HDL from baseline to end of intervention
Changes in total cholesterol | 14 days
  Changes in total cholesterol, measured in mg/dL, from baseline to end of intervention
Changes in LDL cholesterol | 14 days
  Changes in LDL cholesterol, measured in mg/dL, from baseline to end of intervention
Changes in high sensitivity PCR | 14 days
  Changes in high sensitivity PCR, measured in mg/dL, from baseline to end of intervention
Changes in IL-6 | 14 days
  Changes in IL-6, measured in pg/mL, from baseline to end of intervention
Changes in IL-10 | 14 days
  Changes in IL-10, measured in pg/mL, from baseline to end of intervention
Changes in TNFa | 14 days
  Changes in TNFa, measured in pg/mL, from baseline to end of intervention
Changes in adiponectin | 14 days
  Changes in adiponectin, measured in ng/mL, from baseline to end of intervention
Changes in leptin | 14 days
  Changes in leptin, measured in ng/mL, from baseline to end of intervention
Changes in triglycerides | 14 days
  Changes in triglycerides, measured in mg/dL, from baseline to end of intervention
Changes in short chain fatty acids amount in the stool | 14 days
  Changes in short chain fatty acids in the stool, measured in ng/g fecal sample, from baseline to end of intervention
Changes in alkaline phosphatase activity in the stool | 14 days
  Changes in alkaline phosphatase activity in the stool, measured in xx/xx, from baseline to end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ana Faria, PhD, Principal Investigator — Universidade Nova de Lisboa
Locations (1):
- Nova Medical School Universidade Nova de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No